CLINICAL TRIAL: NCT04610697
Title: Cognitive Remediation in Forensic Mental Health Care
Acronym: CRFMHC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TheRoyal
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-04

CONDITIONS: Psychotic Disorders; ADHD; TBI (Traumatic Brain Injury); Aggression; Substance Use Disorders; Violence; Cognitive Dysfunction; Anxiety; Depression; Schizophrenia; Offenders; Antisocial
Keywords: Cognitive Remediation; Cognitive Training; Cognitive Enhancement; Cognitive Rehabilitation; Neuropsychological Rehabilitation; Executive Function; Forensic Mental Health; Forensic Psychology; Forensic Neuropsychology; Forensic Neuroscience; Forensic Rehabilitation; Cognition; Executive Functioning
MeSH Terms: conditions — Psychotic Disorders; Attention Deficit Disorder with Hyperactivity; Brain Injuries, Traumatic; Aggression; Substance-Related Disorders; Cognitive Dysfunction; Anxiety Disorders; Depression; Schizophrenia; Antisocial Personality Disorder | interventions — Cognitive Remediation; Cognitive Training

STUDY DESIGN:
Intervention Model Description: Double blind randomised controlled trial with active control condition. Given the clinically heterogeneous recruitment pool, pseudo-randomization will be employed to match groups on the main diagnosis.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and personnel conducting the assessments will be unaware of group assignment.
  At the halfway mark of recruitment, we will perform preliminary analyses including intention-to-treat liner mixed models. Study staff performing the assessment visits and participants will remain blinded to the study conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Remediation (Experimental): Participants in the cognitive remediation condition will complete computerised exercises followed by bridging discussions delivered using tele-heath.
  More details regarding treatment and control conditions will be provided following study completion to ensure participant blinding.
  Interventions: Behavioral: Cognitive Remediation
- Active control (Active Comparator): Participants in the active control condition will also complete computerised exercises followed by bridging discussions delivered using tele-heath.
  More details regarding treatment and control conditions will be provided following study completion to ensure participant blinding.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Cognitive Remediation — Cognitive Remediation consists of exercises, preferably supported by coaching, aimed at engaging cognitive skills and, as a result, at improving cognition as well as functional and clinical outcomes.
  Other Names: Neuropsychological Rehabilitation; Cognitive Enhancement; Cognitive Rehabilitation
  Arms: Cognitive Remediation
Behavioral: Active Control — Active control condition for cognitive remediation, matched in terms of session modality, number, duration, frequency, and format.
  Arms: Active control

SUMMARY:
Forensic patients often display cognitive deficits, particularly in the domain of executive functions, that represent a challenge to forensic rehabilitation.

One empirically-validated method to train executive functions is cognitive remediation, which consists of cognitive exercises combined with coaching.

This trial investigates whether cognitive remediation can improve cognitive, functional, and clinical outcomes in forensic inpatients.

DETAILED DESCRIPTION:
Forensic patients often display deficits in executive functions, namely difficulties in planning, strategic thinking, problem-solving, and inhibiting inappropriate behavior. Such deficits are transdiagnostic and often underlie behavioral incidents, undermine reintegration into the community, and increase recidivism risk. Despite this, forensic programs usually do not include executive function training.

One approach to train executive functions is cognitive remediation, which consists of behavioral exercises engaging cognitive skills, supported by coaching. In various mental health conditions, cognitive remediation has been repeatedly associated with improvements in cognitive, functional, and clinical outcomes, with small-to-moderate effect sizes. Thus, it should be clarified whether this approach can lead to similar improvements in forensic populations.

In the present trial, we will investigate whether 12 hours over 6 weeks of computerised cognitive remediation administered using tele-health can improve executive functions relative to an active control condition in a sample of 30 forensic inpatients (Aim 1). We will further examine the effect of cognitive remediation (vs. active control) on other variables that are critical for forensic rehabilitation, namely oppositional behaviour, functional capacity, and mental health symptoms (Aim 2). Lastly, we will explore whether any effects persist 12 weeks following cognitive remediation (Aim 3).

Cognitive remediation is an evidence-based inexpensive training method that could be integrated into forensic healthcare practice. In the long term, the expected cognitive, functional, and clinical improvements associated with cognitive remediation have the potential to result in shorter hospitalisations and reduced recidivism rates.

ELIGIBILITY:
Inclusion Criteria:

i1. Age 18 - 55; i2. Ability to read and speak in fluent English; i3. Current status as inpatient on the Forensic Treatment Unit.

Exclusion Criteria:

e1. Intellectual disability; e2. TBI with loss of consciousness followed by known severe neurological sequelae requiring hospitalisation and rehabilitation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Executive Function | within 1 week prior and 1 week after training, as well as at a 12-week follow-up.
  We will measure executive functions using tests from the Cambridge Neuropsychological Test Automated Battery (CANTAB; Sandberg, 2011).

SECONDARY OUTCOMES:
Oppositional Behavior | within 12 weeks before and 12 weeks after training.
  We will measure oppositional behavior using case-manager reports over the 12 weeks preceding and following the study. We will code frequency and severity of behavioral incidents (e.g., verbal and physical aggression) and compliance with rehabilitative interventions.
Functional Capacity | within 1 week prior and 1 week after training, as well as at a 12-week follow-up.
  We will measure perceived functioning in daily life using the Generalized Self-Efficacy Scale (GSES; Schwarzer & Jerusalem, 1995), scored on a scale of 10 to 40, with higher values indicating higher perceived general self-efficacy.
Mental Health Symptoms | within 1 week before and 1 week after training, as well as at a 12-week follow-up.
  We will measure mental health symptoms using the Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM; Evans et al., 2000), scored on a scale of 0 to 136, with greater scores indicating greater psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Pezzoli, PhD, Principal Investigator — UCL and The Royal's Institute of Mental Health Research
Locations (1):
- The Royal's Institute of Mental Health Research, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized datasets will be made available in appropriate online repositories to assist transparency and reproducibility.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be made available upon manuscript preparation (estimated fall 2021).
Access Criteria: Access information will be provided.
URL: https://osf.io/94ukh/